CLINICAL TRIAL: NCT06448429
Title: Evaluating the Integration of Mental Health Care Into the Treatment of Type 1 Diabetes
Brief Title: Testing an Integrated Care Model Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: MQ Mental Health Research (Unknown); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Leslie Johnson, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00007247
Record Dates: First submitted 2024-06-04; First posted 2024-06-07 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Behavioral Health
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Collaborative care group (Experimental): Enrolled participants assigned to the intervention arm will be offered free consultation services with a behavioral health specialist, who is also a licensed clinical social worker.
  Participants randomized into the intervention group will consult with a behavioral health consultant (BHC) one or more times over the intervention period (based on the assessment of the BHC) via phone or Zoom based on the participant's preference.
  The BHC will participate in systematic caseload reviews to facilitate the medical management of depression if indicated.
  Interventions: Other: Usual care; Other: Collaborative care model (CoCM)
- Usual Care (Active Comparator): Participants randomized to the usual care will continue their routine clinical care at the diabetes clinic at Grady.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Usual care — Participants will have the usual diabetes care at the Grady Diabetes Clinic.
  Other Names: Standard of Care (SOC)
Other: Collaborative care model (CoCM) — Collaborative care will include:
  * Care with a behavioral health consultant (BHC)
  * Measurement-based mental health care
  * Systematic caseload reviews
  * Medical management of depression
  The BHC will monitor depression and anxiety severity, promote behavioral change with patients through Behavioral Activation, and support the medical management of depression through participation in caseload reviews (I.e., Mental health care plans for individual patients will be reviewed monthly by a multi-disciplinary T1D clinical team and BHC). Depression treatment initiation (if warranted) by a clinician and engagement in mental health care.
  Other Names: Integrated Care Model
  Arms: Collaborative care group

SUMMARY:
This study aims to test the use of an adapted collaborative care model for improving the health outcomes of adults diagnosed with type 1 diabetes (T1D). The duration of the study is 18 months with 4 study survey points. Participants will fill out an online survey regarding their psychosocial health and chronic disease management behaviors once every six months over the 18 months, and individuals who are randomly assigned to the study intervention will also consult at least once with a behavioral health consultant during the first year (active intervention period).

DETAILED DESCRIPTION:
Type 1 diabetes (T1D) is a lifelong condition that requires consistent monitoring and management, increasing people's risk for common mental disorders that worsen diabetes self-care. Both depression and diabetes can be managed with behavioral interventions, however, they are rarely provided alongside routine diabetes care for people with T1D. In this research study, the investigators aim to evaluate the implementation and effectiveness outcomes of a collaborative care model that uses a Behavioral Health Consultant (BHC) to support lifestyle management among adults with T1D receiving diabetes care at the Grady Diabetes Clinic.

A trained clinical research coordinator will screen interested patients seeking treatment at the Grady Diabetes Center and conduct outreach to individuals who have been identified as having T1D within the Grady Diabetes Center's patient population.

Participants in the intervention group will engage with a behavioral health consultant (BHC) not affiliated with Grady who will work with them to establish personalized health goals and identify ways to manage stress and promote healthy behaviors as means to support their mental and physical health and meet their set goals (i.e., behavioral activation). Each session will be conducted over the telephone or Zoom and last 30-60 minutes, with the number and frequency of meetings established through discussions between the patient and BHC (typically 2-3 sessions for one year). Checklist and summary case reporting templates will be used to track intervention fidelity. The BHC will also participate in ongoing Zoom calls with the multi-disciplinary T1D clinical team at the Grady Diabetes Center once a month to provide updates on patients' behavioral health plans. Transitioning patients from the active intervention will involve discussions with the care team to ensure continued patient support. In cases of active suicidal ideation, the study team will notify the patient's usual diabetes care provider and the individual will be referred to psychiatric services at Grady.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with T1D (based on clinical record diagnosis).

Exclusion Criteria:

* Patients who do not speak English or have reliable telephone access will be excluded. ---
* Individuals with the presence of severe psychiatric illness (PHQ-9≥20) or active suicidal ideation will also be excluded and referred to specialty care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving improvements in PHQ-9 score | Baseline and 12 months
  The proportion of patients achieving improvements in PHQ-9 score [PHQ-9<10] or a ≥50% PHQ-9 score reduction.
Proportion of patients achieving improvement in HbA1c at end of intervention | Baseline and 12 months
  Improvement in HbA1c will be considered as HbA1c<7 or ≥0.5% HbA1c reduction

SECONDARY OUTCOMES:
Generalized anxiety disorder scale score | Baseline and 12 months
  Researchers will use the Generalized anxiety disorder (GAD)-7, a 7-item scale with reporting scores from 0 to 3 on all the questions. It investigates how often the patient has been bothered by seven different symptoms of anxiety during the last two weeks with response options such as: " not at all," " several days '," more than half the days," and " nearly daily " scored as 0, 1, 2, and 3, respectively. The GAD-7 is scored by adding the scores for all 7 items, giving a total score from 0 to 21. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate, and severe anxiety, respectively. Further evaluation is recommended when the score is 10 or greater.
Systolic and diastolic blood pressure (BP) measurements | Baseline and 12 months
  Systolic and diastolic blood pressure (SBP and DBP) will be extracted from participants' medical records.
Low-density lipoprotein (LDL) cholesterol | Baseline and 12 months
  LDL cholesterol data will be extracted from participants' medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Johnson, PhD, MPH, Principal Investigator — Emory University
Locations (1):
- Grady Health System, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers will share deidentified individual participant data that underlie the results reported in published articles, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available beginning 3 months and ending 5 years following article publication.
Access Criteria: Proposals should be directed to lmunoz@emory.edu. To access, the data requesters will sign a data access agreement. Data will be available for 5 years on Emory Dataverse.